CLINICAL TRIAL: NCT05357716
Title: Preliminary Research Evaluation for Ambulatory Leadless Electrocardiogram Recorder Trial
Acronym: PRE-ALERT
Status: Completed | Type: Observational
Sponsor: HelpWear Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1.1
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation; Tachycardia, Supraventricular; Bradyarrhythmia; Ventricular Arrythmia
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Supraventricular; Bradycardia | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Up to 40 patients will be enrolled in Arm A. Subjects will wear the HeartWatch and an Event Recorder for up to 72 hours. Subjects will be asked to document their activities (standing, sitting, walking, exercise, or laying down). Event recorder subjects will collect user-triggered and auto-triggered data.
  Interventions: Device: HeartWatch; Device: Event Recorder
- Arm B: Up to 10 patients will be enrolled in Arm B.Subjects will wear the HeartWatch and Holter monitor for up to 48 hours. Subjects will be asked to document their activities (standing, sitting, walking, exercise, or laying down). Holter subjects will record diary information on their activities and any relevant symptoms.
  Interventions: Device: HeartWatch; Device: Holter Monitor

INTERVENTIONS:
Device: HeartWatch — The HeartWatch arm band provides continuous, high-quality single lead electrocardiograph (ECG) data in a variety of environments. The ECG data is transmitted via Bluetooth and stored on the user's smartphone. It is then uploaded to the cloud for subsequent analysis using either a commercial ECG software package or a customized software package from HelpWear.
Device: Event Recorder — A standard 1 or 2-lead Sirona Event Recorder will be used to collect high-resolution data. Subjects will be asked to wear the clinical monitor for at least 48 hours and no longer than 84 hours. ECG signals will be continuously collected as long as the skin patches are attached to the skin and the recorder is properly connected to the wires.
  Groups: Arm A
Device: Holter Monitor — A standard 5-lead SEER Holter will be used to collect 3-channels of high-resolution data. Subjects will be asked to wear the clinical, conventional monitor for at least 36 hours and no longer than 60 hours. During this time ECG signals will be continuously collected.
  Groups: Arm B

SUMMARY:
The clinical study is intended to implement and test the collection and analysis of paired ECG data from the HeartWatch and two comparator devices, an Event Recorder and Holter. The HeartWatch is indicated for extended diagnostic evaluation of patients with transient symptoms of possible cardiac origin such as syncope and palpitations, as well as patients at risk for arrhythmias, but without significant symptoms. While the use of the device itself can be managed by both healthcare professionals and patients, interpretation of the collected data for diagnosis is restricted to healthcare professionals, as the data must be loaded and analyzed separately after recording. Patients indicated for extended ambulatory ECG testing will be approached for participation. Subjects will wear the HeartWatch and an Event Recorder for up to 72 hours or the HeartWatch and Holter monitor for up to 48 hours. Subjects will be asked to document their activities (standing, sitting, walking, exercise, or laying down). Event recorder subjects will collect user-triggered and auto-triggered data, while Holter subjects will record diary information on their activities and any relevant symptoms. Adverse events and user preference for one device versus the other being used in that arm will also be collected from all subjects. Paired ECG data from the HeartWatch and comparator devices is expected to be similar in terms of the events documented and the proportion of data that is clinically interpretable.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age at time of consent
* Clinically-indicated for an ambulatory Event Recorder or Holter monitor
* Able to follow the protocol
* Provision of written-informed consent

Exclusion Criteria:

* Known allergy to any component of the Event Recorder
* Known allergy to any component of the Holter monitor
* Known allergy to any component of the HeartWatch
* Dextrocardia

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to participating clinics for extended ambulatory ECG testing. Subjects referred for extended ambulatory ECG testing will be recruited from the Toronto Heart Centre. Referring physicians will be asked to indicate if longer-term (i.e., Event Recorder) or shorter-term monitoring (i.e., Holter monitor) is desired for a given patient.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Pairing HeartWatch and Event Recorder | Up to 6 months, with 3 months of analysis time (9 months total)
  Can paired user-triggered (tagged) and auto-triggered ECG data from the HeartWatch and Event Recorder be successfully collected?
Pairing HeartWatch and Holter | Up to 6 months, with 3 months of analysis time (9 months total)
  Can paired continuous ECG data from the HeartWatch and Holter monitor be successfully collected?

SECONDARY OUTCOMES:
Body Position and Activity | Up to 6 months, with 3 months of analysis time (9 months total)
  Does body position and activity affect the quality of the HeartWatch, Event Recorder, and Holter data?

OTHER OUTCOMES:
Adverse Events | Up to 6 months, with 3 months of analysis time (9 months total)
  Incidence of adverse events among the HeartWatch and comparator devices and the types of adverse events
User Preferences | Up to 6 months, with 3 months of analysis time (9 months total)
  User preferences of subjects with the HeartWatch versus the comparator devices

CONTACTS AND LOCATIONS:
Locations (1):
- HelpWear Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT05357716/Prot_000.pdf
  • Informed Consent Form (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT05357716/ICF_001.pdf